CLINICAL TRIAL: NCT02964689
Title: Binimetinib, Pemetrexed and Cisplatin, Followed by Maintenance With Binimetinib and Pemetrexed, in Patients With Advanced Non-small Cell Lung Cancer NSCLC With KRAS Mutations. A Multicenter Phase IB Trial.
Brief Title: Binimetinib in Addition to Standard Chemotherapy in KRAS Mutated NSCLC.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 19/16
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Advanced Non-small Cell Lung Cancer; KRAS Gene Mutation; Lung Cancer
Keywords: Advanced non-small cell lung cancer; KRAS mutations; Binimetinib; Pemetrexed; Cisplatin; Phase IB trial
MeSH Terms: conditions — Lung Neoplasms | interventions — binimetinib; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of binimetinib, pemetrexed and cisplatin (Experimental): The trial consists of two parts:
  * Part 1: dose escalation based on the 3+3 design with 2 doses of binimetinib
  * Part 2: expansion cohort at the recommended maximum tolerated dose (MTD) level of binimetinib
  Interventions: Drug: Binimetinib; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Binimetinib — Binimetinib will be administered in combination with pemetrexed and cisplatin (induction therapy), and with pemetrexed only (maintenance therapy), during the first 2 weeks of each cycle. Cycles will be repeated every 21 days.
  Other Names: MEK162
Drug: Pemetrexed — Pemetrexed 500 mg/m2 i.v. is applied on day 1 of each cycle, before cisplatin administration
Drug: Cisplatin — Cisplatin 75 mg/m2 i.v. is applied on day 1 of each induction therapy cycle. The drug must be administered after pemetrexed infusion

SUMMARY:
The aim is to determine the recommended phase 2 dose (RP2D) of binimetinib in combination with pemetrexed and cisplatin, and to demonstrate that the combination is feasible and has preliminary activity in previously untreated patients with advanced NSCLC and documented KRAS mutations.

DETAILED DESCRIPTION:
There is a need for more effective therapies for patients with advanced NSCLC driven by the RAS/MEK/ERK pathway. These tumors are generally aggressive, are almost exclusively of non-squamous histology, and represent the largest group of patients with advanced NSCLC harboring specific driver mutations in Western populations.

Based on recent preclinical and clinical evidence, mitogen-activated protein kinase kinase (MEK)-inhibition plus first-line chemotherapy is a promising new treatment for patients with NSCLC and KRAS [v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog] mutations.

Binimetinib is a medication without marketing authorization. Pemetrexed and cisplatin have marketing authorization in Switzerland and in EU for the treatment of non-small cell lung cancer (NSCLC) and will be administered as standard backbone treatment according to their Swissmedic-approved indication, dose and route of administration. Binimetinib, pemetrexed and cisplatin are IMP in the context of this phase I trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to the Swiss HRA and ICH-GCP regulation before registration and prior to any trial-specific procedure.
* Histologically or cytologically confirmed diagnosis of NSCLC, predominantly non-squamous subtype (adenocarcinoma, large cell carcinoma, NOS).
* Locally advanced or metastatic stage III-IV disease according to the 7th TNM classification, ineligible for curative treatment.
* Presence of KRAS exon 2 or 3 (codon 12, 13 or 61) mutations by local testing (concomitant EGFR and ALK mutations are excluded).
* CT scan showing measurable disease, which is defined as at least one lesion that can be measured in at least one dimension (non-nodal lesions ≥10 mm in longest diameter, lymph nodes ≥15 mm in short axis) according to RECIST 1.1.
* Eligible for cisplatin-based chemotherapy and able to take oral medications.
* WHO performance status 0-1.
* Age from 18 to 75 years.
* Adequate hematological values: hemoglobin ≥ 90 g/L, ANC ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L.
* Adequate hepatic function: total bilirubin ≤ 1.5 x ULN and < 34.2 μmol/L; ALT and alkaline phosphatase ≤ 2.5 x ULN.
* Adequate renal function: calculated creatinine clearance ≥ 60 mL/min, according to the formula of Cockcroft-Gault.
* Adequate cardiac function: left ventricular ejection fraction (LVEF) ≥ 50% as determined by echocardiogram; QTcF interval must be ≤ 480 ms.
* Women with child-bearing potential are using effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and 6 months thereafter. A negative serum pregnancy test before inclusion into the trial is required for all women with child-bearing potential.
* Men agree not to father a child during trial treatment and 6 months thereafter.

Exclusion Criteria:

* NSCLC with any additional small cell carcinoma (SCLC) component by local diagnostic pathology report.
* Meningeosis carcinomatosa, symptomatic or untreated central nervous system (CNS) metastases. Patients with treated, controlled CNS metastases can be enrolled 2 weeks after the end of radiotherapy if asymptomatic (no residual neurologic deficits) and no longer on corticosteroids.
* Previous or concurrent malignancy with the following exceptions:

  * adequately treated basal cell or squamous cell carcinoma of the skin (adequate wound healing is required prior registration),
  * in situ carcinoma of the cervix, treated curatively and without evidence of recurrence for at least 5 years prior registration,
  * superficial bladder cancer, prostate intraepithelial neoplasm, other noninvasive or indolent malignancy, or other solid tumor treated curatively and without evidence of recurrence for at least 5 years prior registration.
* Leptomeningeal disease.
* Concurrent radiotherapy (patients with prior radiotherapy other than for brain metastases ≥ 7 days prior to registration can be enrolled).
* Previous systemic therapy for advanced NSCLC; previous adjuvant or neoadjuvant chemotherapy allowed if last dose was administered at least 6 months ago.
* Major surgery within 3 weeks before registration.
* Concurrent treatment with any other experimental drug or other anticancer therapy.
* Impaired cardiovascular function or clinically severe or uncontrolled cardiovascular diseases, including any of the following:

  * congestive heart failure NYHA III or IV,
  * history of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) < 6 months prior to registration,
  * symptomatic chronic heart failure (G2 or higher), history or current evidence of clinically significant cardiac arrhythmia requiring medication and/or conduction abnormality < 6 months prior to registration except atrial fibrillation and paroxysmal supraventricular tachycardia.
* Uncontrolled arterial hypertension defined as persistent elevation of systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg despite medical treatment.
* History or current evidence of retinal vein occlusion (RVO) or current risk factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyper-viscosity or hypercoagulability syndromes); history of retinal degenerative disease.
* History of Gilbert's syndrome.
* Neuromuscular disorders that are associated with elevated creatine phosphokinase (CPK; e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* Neuropathy (> G1) or hearing impairment/ tinnitus (> G1).
* Impairment of gastrointestinal function or gastrointestinal disease (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
* History of thromboembolic or cerebrovascular events within 6 months prior to registration, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis or pulmonary emboli.
* Known history of acute or chronic pancreatitis.
* History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) within 12 months prior to registration.
* Known positive serology for HIV (human immunodeficiency virus), active hepatitis B, and/or active hepatitis C infection.
* Active infection within 14 days prior to registration.
* Planning on embarking on a new strenuous exercise regimen after first dose of binimetinib (NB: muscular activities, such as strenuous exercise, that can result in significant increases in plasma CPK levels should be avoided while on binimetinib treatment).
* Known lactose intolerance.
* Known hypersensitivity to the trial drugs or hypersensitivity to any other component of the trial treatment, including premedication.
* Any concomitant drugs contraindicated for use with pemetrexed and cisplatin according to the Swissmedic-approved current product information or with binimetinib according to the latest version of the Investigator's Brochure.
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | within 21 days from the first dose
  A DLT is defined as an AE or abnormal laboratory value assessed as at least possibly related to trial treatment (binimetinib in combination with pemetrexed and cisplatin), which occurs ≤ 21 days following the first dose of trial treatment during cycle 1.

SECONDARY OUTCOMES:
Objective response (OR) | at 30 months after start of trial
  OR will include complete and partial responses based on RECIST 1.1 criteria. Best response will be the best result by investigator and RECIST 1.1 in the planned follow-up CT scans.
Progression-free survival (PFS) | at 30 months after start of trial
  PFS will be calculated from registration until documented tumor progression according to RECIST 1.1 or death due to any reason, whichever occurs first.
Overall survival (OS) | at 30 months after start of trial
  OS will be calculated from registration until death due to any reason.
Adverse events (AEs) | at 30 months after start of trial
  AEs will be assessed according to NCI CTCAE V.4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Früh, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (4):
- Switzerland (4):
  - Universitaetsspital Basel, Basel
  - IOSI Ospedale Regionale di Bellinzona e Valli, Bellinzona
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No